CLINICAL TRIAL: NCT00556088
Title: A Phase I Study of LBH589 in Combination With Paclitaxel and Carboplatin +/- Bevacizumab the Treatment of Solid Tumors
Brief Title: LBH589, Paclitaxel, Carboplatin +/- Bevacizumab for Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Howard A. Burris, III, M.D., Sarah Cannon Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 121
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-12

CONDITIONS: Solid Tumors
Keywords: LBH589; Phase I; Solid Tumors; Paclitaxel; Carboplatin; Bevacizumab; Dose escalation
MeSH Terms: interventions — Panobinostat; Paclitaxel; Carboplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Part 1 (Experimental): Part I Phase I dose escalation trial. LBH589 will be administered orally on Monday and Thursday or Tuesday and Friday each week (twice weekly). Paclitaxel and carboplatin will be administered intravenously every 21 days.
  Part II LBH589, paclitaxel, and carboplatin dosing will be determined in the first phase of this study (Phase I). The drug dosages to be administered will be reduced one level from the determined Maximum Tolerated Dose (MTD). In addition, bevacizumab 15 mg/kg will be added to the second portion of this trial.
  Interventions: Drug: LBH589, Paclitaxel, Carboplatin, Bevacizumab

INTERVENTIONS:
Drug: LBH589, Paclitaxel, Carboplatin, Bevacizumab — LBH589 will be administered orally twice weekly. Paclitaxel and carboplatin will be administered intravenously every 21 days.
  Once the MTD is established, drug dosages will be adjusted downward by one dose level and bevacizumab 15mg/kg intravenously every 3 weeks will be administered to a subset of patients with non-small cell lung cancer.

SUMMARY:
This phase I protocol will evaluate the safety and tolerability of the combination of LBH589 and paclitaxel/carboplatin. The combination of LBH589, paclitaxel/carboplatin, and bevacizumab will also be evaluated for tolerability and preliminary antitumor activity in a subset of patients with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented metastatic or locally advanced, incurable malignancy for which paclitaxel and carboplatin is clinically appropriate for example, non-small cell lung, breast, ovarian, head and neck cancer, and carcinoma of unknown primary.
2. Male or female patients aged >= 18 years old.
3. Maximum of 3 prior regimens in a metastatic setting allowed and may include other targeted agents, immunotherapy and chemotherapy.
4. Measurable disease by RECIST criteria.
5. ECOG PS 0 or 1.
6. Laboratory values as follows:

   ANC >= 1500/μL Hgb >= 9 g/dL Platelets >= 100,000/uL Bilirubin <= upper limit normal (ULN) AST/SGOT and ALT/SGPT <= 2.5 x ULN or <= 5.0 x ULN in patients with liver metastases Creatinine <= 2.0 mg/dL Or 24-hour Creatinine Clearance >= 50 ml/min Albumin >= 3 g/dL Potassium >= lower limit normal (LLN) Phosphorous >= LLN Calcium >= LLN Magnesium >= LLN PT/INR and PTT <= 1.5 x ULN
7. Peripheral neuropathy < grade 1.
8. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment.
9. Life expectancy > 12 weeks.
10. Accessible for treatment and follow-up.
11. All patients must be able to understand the nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
2. Impaired cardiac function including any of the following:

   * Screening ECG with a QTc > 450 msec.
   * Congenital long QT syndrome.
   * History of sustained ventricular tachycardia.
   * Any history of ventricular fibrillation or torsades de pointes.
   * Bradycardia defined as heart rate < 50 beats per minutes. Patients wit a pacemaker and heart rate >= 50 beats per minute are eligible.
   * Myocardial infarction or unstable angina within 6 months of study entry.
   * Congestive heart failure (NY Heart Association class III or IV [See Appendix B]).
   * Right bundle branch block and left anterior hemiblock (bifasicular block).
   * Atrial fibrillation or flutter.
3. Uncontrolled hypertension (systolic blood pressure [BP] 160 or diastolic BP >95mm Hg) or uncontrolled cardiac arrhythmias.
4. Active CNS disease, including meningeal metastases.
5. Known diagnosis of human immunodeficiency virus (HIV) infection.
6. Unresolved diarrhea > CTCAE grade 1.
7. Chemotherapy, investigational drug therapy, major surgery < 4 weeks prior to starting study drug or patients that have not recovered from side effects of previous therapy.
8. Patient is < 5 years free of another primary malignancy except if the other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
9. Concomitant use of any anti-cancer therapy or radiation therapy.
10. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP) not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days of the first administration of oral LBH589.
11. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom.
12. Patients with gastrointestinal (GI) tract disease, causing the inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
13. Other concurrent severe, uncontrolled infection or intercurrent illness, including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
14. Patients with uncontrolled coagulopathy.
15. Abnormal thyroid function (TSH or free T4) detected at screening.Patients with known hypothyroidism who are stable on thyroid replacement are eligible.

Exclusion Criteria (Part II portion)

1. Patients with tumor types other than advanced non-small cell lung cancer and patients with squamous cell histology non-small cell lung cancer.
2. Patients who have had a major surgical procedure (not including mediastinoscopy), open biopsy, or significant traumatic injury within 6--8 weeks of beginning bevacizumab. Fine needle aspiration, core biopsy, mediastinoscopy or other minor surgical procedure within 7 days of beginning bevacizumab.
3. Patients receiving full-dose oral or parenteral anticoagulation. Patients receiving thrombolytic therapy within 10 days of starting bevacizumab are also ineligible. Patients may receive anticoagulation therapy, (1 mg coumadin daily) for port clot prophylaxis.
4. Patients with serious non-healing wound, ulcer, or bone fracture.
5. Patients with evidence of bleeding diathesis or coagulopathy.
6. Patients with history of hemoptysis (defined as bright red blood of ½ teaspoon or more per episode) within 3 months prior to study enrollment.
7. History of myocardial infarction or unstable angina within 6 months of first bevacizumab dose.
8. Patients with proteinuria at screening for as demonstrated by either:

   a. Urine protein creatinine (UPC) ration >1.0 at screening OR b. Urine dipstick for proteinuria > 2+ (patients discovered to have > 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate < 1 g of protein in 24 hours to be eligible.
9. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to beginning bevacizumab.
10. History of stroke or transient ischemic attack within 6 months prior to first bevacizumab dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Determine the maximally tolerated doses and dose limiting toxicities of LBH589 in combination with paclitaxel and carboplatin. Preliminary anti-tumor activity will also be assessed. | 18 months

SECONDARY OUTCOMES:
Determine the tolerability and preliminary efficacy in a subset of patients with non-small cell lung cancer. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Burris, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States